CLINICAL TRIAL: NCT04576117
Title: A Phase 3 Study of Selumetinib (NSC# 748727) or Selumetinib in Combination With Vinblastine for Non-NF1, Non-TSC Patients With Recurrent or Progressive Low-Grade Gliomas (LGGs) Lacking BRAFV600E or IDH1 Mutations
Brief Title: A Study to Compare Treatment With the Drug Selumetinib Alone Versus Selumetinib and Vinblastine in Patients With Recurrent or Progressive Low-Grade Glioma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-07549; NCI-2020-07549 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACNS1931 (Other: Children's Oncology Group); ACNS1931 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2020-10-03; First posted 2020-10-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Recurrent Low Grade Astrocytoma; Recurrent WHO Grade 2 Glioma; Refractory Low Grade Astrocytoma; Refractory Low Grade Glioma; Refractory WHO Grade 1 Glioma
MeSH Terms: interventions — Specimen Handling; Magnetic Resonance Spectroscopy; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efficacy Phase Arm II (selumetinib) (Active Comparator): Patients receive selumetinib sulfate PO BID on days 1-28. Treatment repeats every 28 days for up to 27 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo MRI throughout the trial. Patients also undergo blood sample collection during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Selumetinib Sulfate
- Feasibility & Efficacy Phase Arm I (selumetinib, vinblastine) (Experimental): Patients receive vinblastine sulfate IV over 1 minute or IV infusion on days 1, 8, 15, and 22 and selumetinib sulfate PO BID on days 1-28. Treatment repeats every 28 days. Patients receive selumetinib and vinblastine for a total duration of 17 cycles followed by 10 additional cycles of selumetinib alone in the absence of disease progression or unacceptable toxicity. Patients undergo MRI throughout the trial. Patients also undergo blood sample collection during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Selumetinib Sulfate; Drug: Vinblastine Sulfate

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Selumetinib Sulfate — Given PO
  Other Names: AZD-6244 Hydrogen Sulfate; AZD6244 Hydrogen Sulfate; AZD6244 Hydrogen Sulphate; Koselugo; Selumetinib Sulphate
Drug: Vinblastine Sulfate — Given IV
  Other Names: 29060 LE; 29060-LE; Exal; Velban; Velbe; Velsar; VINCALEUKOBLASTINE
  Arms: Feasibility & Efficacy Phase Arm I (selumetinib, vinblastine)

SUMMARY:
This phase III trial investigates the best dose of vinblastine in combination with selumetinib and the benefit of adding vinblastine to selumetinib compared to selumetinib alone in treating children and young adults with low-grade glioma (a common type of brain cancer) that has come back after prior treatment (recurrent) or does not respond to therapy (progressive). Selumetinib is a drug that works by blocking a protein that lets tumor cells grow without stopping. Vinblastine blocks cell growth by stopping cell division and may kill cancer cells. Giving selumetinib in combination with vinblastine may work better than selumetinib alone in treating recurrent or progressive low-grade glioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose/recommended phase 2 dose (MTD/RP2D) of selumetinib sulfate (selumetinib) + vinblastine sulfate (vinblastine) for children with progressive or recurrent low-grade gliomas (LGGs).

II. To determine if selumetinib + vinblastine will lead to improved event-free survival (EFS) outcome compared with selumetinib alone for children with progressive or recurrent LGGs.

SECONDARY OBJECTIVES:

I. To estimate the objective response rates and overall survival associated with treatment with selumetinib + vinblastine versus single-agent selumetinib.

II. To estimate the difference in EFS and response rate between patients with BRAF rearranged LGG and patients with non-BRAF rearranged LGG after treatment with selumetinib + vinblastine versus single-agent selumetinib.

III. To evaluate toxicities associated with selumetinib + vinblastine and single-agent selumetinib for children with progressive or recurrent LGGs.

IV. To compare the quality of life among patients treated with selumetinib + vinblastine and single-agent selumetinib.

V. To examine the vision outcomes among patients with optic pathway gliomas (OPGs) treated with selumetinib + vinblastine and single-agent selumetinib.

EXPLORATORY OBJECTIVE:

I. To obtain paired blood and tumor specimens for future biology studies, including studies to correlate genomic drivers to response.

OUTLINE: This is a dose-escalation feasibility study of vinblastine sulfate in combination with selumetinib, followed by a randomized efficacy study. Patients in the feasibility study are assigned to Arm I, while patients in the efficacy study are randomized to Arm I or Arm II.

ARM I: Patients receive vinblastine sulfate intravenously (IV) over 1 minute or IV infusion on days 1, 8, 15, and 22 and selumetinib sulfate orally (PO) twice daily (BID) on days 1-28. Treatment repeats every 28 days. Patients receive selumetinib and vinblastine for a total duration of 17 cycles followed by 10 additional cycles of selumetinib alone in the absence of disease progression or unacceptable toxicity. Patients undergo magnetic resonance imaging (MRI) throughout the trial. Patients also undergo blood sample collection during screening and on study.

ARM II: Patients receive selumetinib sulfate PO BID on days 1-28. Treatment repeats every 28 days for up to 27 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo MRI throughout the trial. Patients also undergo blood sample collection during screening and on study.

After completion of study treatment, patients are followed up every 3 months for year 1, every 6 months for years 2-3, and annually for years 4-5.

ELIGIBILITY:
Inclusion Criteria:

* Feasibility phase: patients must be >= 2 years and =< 21 years of age at the time of enrollment
* Efficacy phase: patients must be >= 2 years and =< 25 years of age at the time of enrollment

  * All patients > 21 years of age at the time of enrollment must have had initial diagnosis of low-grade glioma by 21 years of age
* Patients must have a body surface area (BSA) of >= 0.5 m^2 at enrollment
* Patients must have eligibility confirmed by rapid central pathology and central molecular screening reviews performed on APEC14B1

  * Non-neurofibromatosis type 1 (non-NF1), non-tuberous sclerosis complex (non-TSC) low-grade glioma (LGG) without a BRAFV600E or IDH1 mutation
  * Patients must have progressive or recurrent LGG. Note: Biopsy may be at either initial diagnosis or recurrence
  * Patients must have measurable disease, defined as having a two-dimensional measurable tumor volume of >= 1 cm^2

    * Tumor size will be measured to include both solid and cystic components of the tumor (whether or not tumor is enhancing) + fluid attenuated inversion recovery (FLAIR) signal
  * Eligible histologies will include all tumors considered low-grade glioma or low-grade astrocytoma (World Health Organization [WHO] grade 1 and II) by the WHO Classification of Tumors of the Central Nervous System - 4th Edition Revised, with the exception of subependymal giant cell astrocytoma
  * Patients with metastatic disease or multiple independent primary LGGs are eligible
* Patients must be progressive or recurrent after having been treated with at least one prior tumor-directed therapy before enrollment
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study

  * Myelosuppressive chemotherapy: Must not have received within 2 weeks of entry onto this study (4 weeks if prior nitrosourea);
  * Biologic (anti-neoplastic agent): At least 7 days since the completion of therapy with a biologic agent;
  * Radiation therapy (RT): >= 2 weeks (wks) for local palliative RT (small port); >= 6 months must have elapsed if prior craniospinal RT or if >= 50% radiation of pelvis; >= 6 wks must have elapsed if other substantial bone marrow (BM) radiation;
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to =< grade 1;
  * MEK inhibitor or vinblastine: Must not have received treatment with a MEK inhibitor or vinblastine within 6 months of study enrollment
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^ 2 or a serum creatinine based on age/sex as follows (within 7 days prior to enrollment):

  * 2 to < 6 years: 0.8 mg/dL (male) 0.8 mg/dL (female)
  * 6 to < 10 years: 1 mg/dL (male) 1 mg/dL (female)
  * 10 to < 13 years: 1.2 mg/dL (male) 1.2 mg/dL (female)
  * 13 to < 16 years: 1.5 mg/dL (male) 1.4 mg/dL (female)
  * >= 16 years: 1.7 mg/dL (male) 1.4 mg/dL (female)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age (within 7 days prior to enrollment) (children with a diagnosis of Gilbert's syndrome will be allowed on study regardless of their total and indirect [unconjugated] bilirubin levels as long as their direct [conjugated] bilirubin is < 3.1 mg/dL)
* Serum glutamic pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L (within 7 days prior to enrollment)

  * Note: For the purpose of this study, the ULN for SGPT (ALT) has been set to the value of 45 U/L
* Albumin >= 2 g/L (within 7 days prior to enrollment)
* Left ventricular ejection fraction (LVEF) >= 53% (or institutional normal; if the LVEF result is given as a range of values, then the upper value of the range will be used) by echocardiogram (within 4 weeks prior to enrollment)
* Corrected QT interval (QTc interval) =< 450 msec by electrocardiogram (EKG) (within 4 weeks prior to enrollment)
* Absolute neutrophil count >= 1,000/uL (unsupported) (within 7 days prior to enrollment)
* Platelets >= 100,000/uL (unsupported) (within 7 days prior to enrollment)
* Hemoglobin >= 8 g/dL (may be supported) (within 7 days prior to enrollment)
* Patients with a known seizure disorder should be stable and should not have experienced a significant increase in seizure frequency within 2 weeks prior to enrollment
* Stable neurological examination for >= 1 week
* HYPERTENSION:

  * Patients 2-17 years of age must have a blood pressure that is =< 95th percentile for age, height, and sex at the time of enrollment (with or without the use of anti-hypertensive medications);
  * Patients >= 18 years of age must have a blood pressure =< 130/80 mmHg at the time of enrollment (with or without the use of anti-hypertensive medications)
  * Note for patients of all ages: Adequate blood pressure can be achieved using medication for the treatment of hypertension
* All patients must have ophthalmology toxicity assessments performed within 4 weeks prior to enrollment
* For all patients, an MRI of the brain (with orbital cuts for optic pathway tumors) and/or spine (depending on the site[s] of primary disease) with and without contrast must be performed within 4 weeks prior to enrollment

  * Note: If surgical resection or biopsy is performed at the time of progression or recurrence, a post-operative MRI is required
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1, or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Patients must have the ability to swallow whole capsules

Exclusion Criteria:

* Prior therapy with vinblastine and/or a MEK inhibitor is permitted, with the following exceptions:

  * Patients must not have had progressive disease while on therapy with vinblastine or a MEK inhibitor;
  * Patients must not have discontinued vinblastine or selumetinib due to toxicity
* Patients with a concurrent malignancy or history of treatment (other than surgery) for another tumor within the last year are ineligible
* Patients with diffuse intrinsic pontine tumors as seen on MRI (> 2/3 of pons involvement on imaging) are not eligible even if biopsy reveals grade I/II histology
* Patients may not be receiving any other investigational agents
* Patients must not have known hypersensitivity to selumetinib, vinblastine, or similar compounds
* CYP3A4 agents: Patients must not have received fluconazole or drugs that are strong inducers or inhibitors of CYP3A4 within 7 days prior to study enrollment
* Patients with any serious medical or psychiatric illness/condition, including substance use disorders or ophthalmological conditions, likely in the judgment of the investigator to interfere or limit compliance with study requirements/treatment
* Patients who, in the opinion of the investigator, are not able to comply with the study procedures are not eligible
* PRE-EXISTING CONDITIONS (CARDIAC):

  * Known genetic disorder that increases risk for coronary artery disease. Note: The presence of dyslipidemia in a family with a history of myocardial infarction is not in itself an exclusion unless there is a known genetic disorder documented;

    * Symptomatic heart failure
    * New York Heart Association (NYHA) class II-IV prior or current cardiomyopathy
    * Severe valvular heart disease
    * History of atrial fibrillation
* PRE-EXISTING CONDITIONS (OPHTHALMOLOGIC CONDITIONS):

  * Current or past history of central serous retinopathy
  * Current or past history of retinal vein occlusion or retinal detachment
  * Patients with uncontrolled glaucoma

    * If checking pressure is clinically indicated, patients with intraocular pressure (IOP) > 22 mmHg or upper limit of normal (ULN) adjusted by age are not eligible
* Any multivitamin containing vitamin E must be stopped prior to study enrollment even if it contains less than 100% of the daily recommended dosing for vitamin E
* Surgery within 2 weeks prior to enrollment, with the exception of a surgical biopsy, placement of a vascular access device or cerebrospinal fluid (CSF) diverting procedure such as endoscopic third ventriculostomy (ETV) and ventriculoperitoneal (VP) shunt

  * Note: Patients must have healed from any prior surgery
* Patients who have an uncontrolled infection are not eligible
* Female patients who are pregnant are not eligible since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential
* Lactating females who plan to breastfeed their infants
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation and for 12 weeks after stopping study therapy are not eligible

  * Note: Women of child-bearing potential and males with sexual partners who are pregnant or who could become pregnant (i.e., women of child-bearing potential) should use effective methods of contraception for the duration of the study and for 12 weeks after stopping study therapy to avoid pregnancy and/or potential adverse effects on the developing embryo
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-02-16 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose/recommended phase II dose (MTD/RP2D) of selumetinib and vinblastine combination (feasibility) | 1 month post enrollment
  The MTD is empirically defined as the highest dose level at which 6 patients have been treated with at most one patient experiencing a dose-limiting toxicity (DLT) and the next higher dose level has been determined to be too toxic.
Event-free survival (efficacy) | Up to 5 years after enrollment
  Will use Kaplan-Meier (KM) methods and stratified log-rank tests to estimate EFS per arm and compare the EFS outcome between the two arms to assess difference in efficacy. EFS is defined as the interval from randomization to the first occurrence of clinical or radiographic disease progression, disease recurrence, subsequent malignant neoplasm, or death from any cause. Patients who are event-free will be censored at the time of last follow-up.

SECONDARY OUTCOMES:
Radiographic tumor response rate (efficacy) | Up to 2 years after enrollment
  Will summarize the radiologic response rates (complete response [CR] or partial response [PR] per arm and test for a difference between the 2 arms using an exact binomial test. PR is defined as greater than or equal to 50% reduction in target lesion size by bi-dimensional measurement on T2/FLAIR, as compared with the baseline measurements, on a stable or decreasing dose of corticosteroids, accompanied by a stable or improving neurologic examination, and maintained for at least 8 weeks. CR must also be sustained for at least 8 weeks and requires complete disappearance of the target lesion on T2/FLAIR imaging (if enhancement had been present, it must have resolved completely); No new lesions, no new T2/FLAIR abnormalities, and no new or increased enhancement; Patients must be off corticosteroids or only on physiological replacement doses; and Patients should be stable or improved clinically.
Overall survival (OS) (efficacy) | Up to 5 years after enrollment
  Will use the KM methods to estimate OS for each treatment arm and use stratified log-rank tests to determine whether there is a difference in OS between the 2 arms. OS is defined as the interval from randomization to death from any cause or to the time of last follow-up for patients who are alive at the time of analysis
EFS by BRAF Status | Up to 5 years after enrollment
  Will use KM methods to estimate the difference in EFS and between patients with BRAF rearranged LGG and patients with non-BRAF rearranged LGG after treatment with selumetinib + vinblastine versus single-agent selumetinib. EFS is defined as the interval from randomization to the first occurrence of clinical or radiographic disease progression, disease recurrence, subsequent malignant neoplasm, or death from any cause. Patients who are event-free will be censored at the time of last follow-up
Incidence of adverse events (feasibility) | Up to 5 years
  Toxicities will be summarized by dose level and by attribution to vinblastine versus selumetinib during the feasibility component.
Incidence of adverse events (efficacy) | Up to 5 years
  Reported toxicities will be summarized per arm for the efficacy component.
Quality of life (QOL) | Baseline to cycle 7 day 1
  Will use 2-sample 2-sided t-tests to compare the change from baseline in the PedsQL™ Generic Module Total Scale Score between the two treatment arms at Cycle 7 Day 1 for both patient and parent-proxy report.
Visual outcome comparison | 12 months after enrollment
  Will use an exact binomial test to compare the difference in the proportion of subjects in each arm that show improvement in visual acuity per Teller Acuity assessment after 12 months of treatment using a 1-sided test with 10% type 1 error.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Bowers, Principal Investigator — Children's Oncology Group
Locations (101):
- United States (91):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Maine Children's Cancer Program, Scarborough, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (10):
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (2):
  • Informed Consent Form: PACNS1931_A02ConsentPartA(SafetyPhase)(Redacted).pdf (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT04576117/ICF_001.pdf
  • Informed Consent Form: PACNS1931_A02ConsentPartB(EfficacyPhase)(Redacted).pdf (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT04576117/ICF_000.pdf